CLINICAL TRIAL: NCT04936217
Title: Long-term Evaluation of the Efficacy and Safety of a Continent Cutaneous Urinary Diversion in Spinal Cord Injury Patients
Brief Title: Efficacy and Safety of a Continent Cutaneous Urinary Diversion in Spinal Cord Injury Patients
Acronym: ELESDUCCBM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local 2019/SD-01
Record Dates: First submitted 2021-06-18; First posted 2021-06-23 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Spinal Cord Injuries; Urinary Diversion; Neurogenic Bladder
Keywords: intermittent catheterization; Mitrofanoff; Yang-Monti
MeSH Terms: conditions — Spinal Cord Injuries; Urinary Bladder, Neurogenic | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients operated for Continent Cutaneous Urinary Diversion, April 2004 - October 2017: The study focuses of a population of 70 patients operated between April 2004 and October 2017 au Nîmes University Hospital for Cutaneous Urinary Diversion.
  Interventions: Other: Data collection; Other: Interview using a validated questionnaire

INTERVENTIONS:
Other: Data collection — For each patient, the following data will be collected and analyzed: age at operation, sex, Body Mass Index (BMI), ASA score, ASIA score, type of bladder dysfunction assessed by urodynamic evaluation, urinary abnormalities assessed by morphological examination (ultrasound and / or computed tomography) and cystoscopy, creatinine clearance, operative indications, initial mictional mode, surgical assembly, immediate and later complications.
Other: Interview using a validated questionnaire — A telephone survey will be conducted by means of a questionnaire in order to evaluate the patient's quality of life.

SUMMARY:
Continent Cutaneous Urinary Deviation (CUD), using the Mitrofanoff, Yang-Monti or Casale principle, is offered to patients with neurological diseases who are unable to perform intermittent catheterisation through the native urethra due to upper limb disability.

There is very little data in the literature examining the long-term efficacy and complications of this technique. The main objective of this study is to evaluate the effectiveness of long-term CUDs in spinal cord injury patients. The secondary objectives are to evaluate the surgical complications and the impact on the patient's quality of life.

For each patient, several data will be collected and analyzed: age at operation, sex, Body Mass Index (BMI), ASA score, ASIA score, type of bladder dysfunction assessed by urodynamic evaluation, urinary abnormalities assessed by morphological examination (ultrasound and / or computed tomography) and cystoscopy, creatinine clearance, operative indications, initial mictional mode, surgical assembly and any immediate or late complications. In a second stage, a questionnaire survey will be conducted by telephone.

ELIGIBILITY:
Inclusion Criteria:

Specific inclusion criteria for the study :

* no history of continuous cystostomy in another centre
* a follow-up > 24 months,
* a continent cutaneous urinary diversion for a spinal cord injury.

General inclusion criteria :

* Patient affiliated to or beneficiary of a health insurance scheme.
* Adult patient (≥18 years of age) and under 85 years of age.

Exclusion Criteria:

* Criteria for non-inclusion specific to the study :
* All urinary incontinence outside of medullary waiting period.
* A history of continuous cystostomy in another centre.
* A follow-up of less than 24 months,
* a continent cutaneous urinary diversion for a neurological pathology other than spinal cord injury.

General criteria for non-inclusion :

* Patient in a period of exclusion determined by another study.
* Patient for whom it is impossible to give enlightened information.
* Patient under legal protection, guardianship or curatorship.
* Patient unable to express consent

Min Age: 17 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients who have suffered a spinal cord injury, operated on between April 2004 and October 2017 at Nîmes University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of continent cutaneous urinary derivation: catheterisation. | 3 -16 years after their operation
  The minimum frequency of urinary catheterisation in spinal injured patients equipped with a continent cutaneous urinary derivation will be recorded.
Efficacy of continent cutaneous urinary derivation:leakage | 3 -16 years after their operation
  Absence of leakage through the cystostomy in spinal injured patients equipped with a continent cutaneous urinary derivation will be recorded.

SECONDARY OUTCOMES:
Surgical complications and impact on the patient's quality of life: Age at start of care | 3 -16 years after their operation
  The patient's age will be noted at the start of care
Surgical complications and impact on the patient's quality of life: Sex | 3 -16 years after their operation
  The patient's sex will be noted at the start of care
Surgical complications and impact on the patient's quality of life: Body Mass Index | 3 -16 years after their operation
  The patient's Body Mass Index will be noted at the start of care
Surgical complications and impact on the patient's quality of life: ASA score | 3 -16 years after their operation
  The ASA Physical Status Classification System is used to assess and communicate a patient's pre-anesthesia medical comorbidities. The classification system alone does not predict the perioperative risks, but used with other factors (eg, type of surgery, frailty, level of deconditioning) it can be helpful in predicting perioperative risks.
  ASA I = A normal healthy patient ASA II = A patient with mild systemic disease ASA III = A patient with severe systemic disease ASA IV = A patient with severe systemic disease that is a constant threat to life ASA V = A moribund patient who is not expected to survive without the operation ASA VI = A declared brain-dead patient whose organs are being removed for donor purposes
Surgical complications and impact on the patient's quality of life: ASIA score | 3 -16 years after their operation
  The ASIA (American Spinal Injury Association) assessment is the gold standard for assessing and documenting sensory and motor impairments after Spinal Cord Injury. The score ranges from A to E as follows:
  A = Complete injury. No motor or sensory function is preserved in the sacral segments S4 or S5.
  B = Sensory incomplete. Sensory but not motor function is preserved below the level of injury, including the sacral segments.
  C = Motor incomplete. Motor function is preserved below the level of injury, and more than half of muscles tested below the level of injury have a muscle grade less than 3 (see muscle strength scores table).
  D = Motor incomplete. Motor function is preserved below the level of injury and at least half of the key muscles below the neurological level have a muscle grade of 3 or more.
  E = Normal. No motor or sensory deficits, but deficits existed in the past. This score will be used to evaluate the patient at the start of care.
Surgical complications and impact on the patient's quality of life: Bladder dysfunction | 3 -16 years after their operation
  The type of bladder dysfunction will be evaluated by urodynamic evaluation
Surgical complications and impact on the patient's quality of life: urinary tract anomalies evaluated via a morphological examination. | 3 -16 years after their operation
  Urinary tract anomalies will be evaluated via a morphological examination (using ultrasound and / or tomodensitometry).
Surgical complications and impact on the patient's quality of life: cytometry | 3 -16 years after their operation
  Urinary tract anomalies will be evaluated via cytometry
Surgical complications and impact on the patient's quality of life: creatinine clearance | 3 -16 years after their operation
  Urinary tract anomalies will be evaluated according to the patient's creatinine clearance
Surgical complications and impact on the patient's quality of life: operative indications | 3 -16 years after their operation
  The indications for the initial surgery will be recorded.
Surgical complications and impact on the patient's quality of life: mictional mode | 3 -16 years after their operation
  The patient's initial mictional mode will be recorded.
Surgical complications and impact on the patient's quality of life: surgical set-up | 3 -16 years after their operation
  The patient's surgical set-up will be recorded.
Surgical complications and impact on the patient's quality of life: immediate or later complications | 3 -16 years after their operation
  All immediate or later complications will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France